CLINICAL TRIAL: NCT04105426
Title: A Phase-II Clinical Trial on the Effectiveness of Antioxidant Supplementation in Idiopathic Tinnitus Patients
Brief Title: A Study on the Effectiveness of Antioxidant Supplementation in Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Anna Petridou, Dietitian-Nutritionist, M.Med.Sci, PhD candidate, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4354
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidants (Active Comparator): This arm of patients received one multivitamin and multimineral tablet with 500 mg grape seed extract once a day and one tablet of alpha-lipoic acid (300 mg ALA) twice a day for 3 months.
  Interventions: Dietary Supplement: Antioxidants
- Placebo (Placebo Comparator): This arm of patients received placebo for 3 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidants — one multivitamin and multimineral tablet with 500 mg grape seed extract once a day and one tablet of alpha-lipoic acid (300 mg ALA) twice a day for 3 months.
  Arms: Antioxidants
Dietary Supplement: Placebo — one placebo tablet three times per day for 3 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of antioxidant supplementation in idiopathic tinnitus patients.

To investigate this, a double-blind, randomized, and placebo-controlled clinical trial was conducted to assess the impact of a multivitamin-multimineral supplement with phytochemicals combined with a-lipoic acid supplements on serum oxidative stress, serum antioxidant capacity and tinnitus parameters in patients with idiopathic tinnitus.

Subjective, idiopathic, non-pulsatile tinnitus ("tinnitus") is perception of sound without the presence of an external acoustic stimulus. Causes of idiopathic tinnitus remain unknown and the pathological mechanisms are not fully understood. Currently, effective therapies for tinnitus remain limited. Previous research has demonstrated that oxidative stress is possibly involved in the pathogenesis of idiopathic tinnitus and some studies have shown beneficial effects of antioxidant therapy in tinnitus patients. Moreover, many studies have shown the beneficial effect of antioxidant supplementation on the reduction of oxidative stress and the increase of endogenous antioxidant enzymes and antioxidant capacity.

Seventy patients with idiopathic tinnitus were enrolled based on certain inclusion and exclusion criteria. Subsequently, they were informed regarding the aims, methods, anticipated benefits, and potential hazards of the study, and were provided with the information leaflet of the study. Each patient who agreed to take part in the study, signed an informed consent form, a copy of which was given to them.

Participants were allocated to either antioxidant or placebo group. Randomisation was conducted by someone who was not involved in the study and blinding was strictly maintained to researchers and participants.

The antioxidant group received one multivitamin and multimineral tablet with grape seed extract once a day together with one tablet of alpha-lipoic acid twice a day, whereas the placebo group received identical placebo tablets. Supplements were kindly donated by Lamberts. The intervention lasted 3 months. Both groups kept their usual medical treatment and their diet and exercise habits stable during the intervention.

Patients were assessed after randomisation according to the following tools:

* Medical history
* Audiometric and Tinnitus assessment: Basic audiometric tests, pitch match, loudness match, minimum masking level (MML)
* Tinnitus questionnaires: Tinnitus Handicap Inventory (THI), Tinnitus Functional Index (TFI) and Visual Analogue Scale (VAS)
* anthropometrics: body weight , height, Body Mass Index, waist and hip circumferences
* Nutrition and physical activity evaluation
* Adherence to the Mediterranean dietary pattern (MedDietScore)
* Psychological assessment
* Biochemical measurements: Complete blood count, lipid profile, glucose, electrolytes, liver enzymes, thyroid hormones
* Vitamin laboratory tests
* Oxidative stress assessment in serum samples: Total Antioxidant Capacity (TAC), Superoxide Dismutase (SOD) activity and Oxidized LDL are quantified.

Compliance and any side effects were checked with a weekly telephone contact with the patients. The consumption of tablets was checked with a diary completed by patients. At the end of the intervention, all baseline parameters were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-75 years old
* Unilateral or bilateral chronic idiopathic persistent tinnitus of at least 6 months' duration
* Tinnitus Handicap Inventory score rated ≥ 4 at baseline
* With a normal audiogram or up to medium-grade neurosensory hearing loss.
* Tinnitus maskable (by noise masking) with noise at least 5 decibel
* Childbearing age with a negative pregnancy test at eligibility and baseline assessment
* Stable medication during the whole period of the 3-month intervention
* Willing and able to attend the on-study visits
* Able to read and understand the relevant study documents and rating scales and follow investigator instructions during audiologic measurements

Exclusion Criteria:

* Tinnitus following acute acoustic trauma, sudden deafness or traumatic head or neck injury
* Intermittent tinnitus
* Meniere's Disease, otosclerosis, acute or chronic otitis media
* Head and neck radiotherapy
* Active GI disease; active malignant diseases; autoimmune diseases; cardiovascular disease; renal or hepatic disorders; haemorrhagic diathesis
* Intake of anticoagulants; ototoxic medications; tinnitus-inducing medication (e.g. aminoglycosides, chemotherapeutics, loop diuretics, high doses of aspirin or quinine)
* Psychiatric disorders
* Unregulated diabetes mellitus, hypertension or thyroid disease
* Alcohol or drug abuse
* Vitamin or inorganic supplements, vegan or macrobiotic diet before and during the trial
* Pregnancy, lactation

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Tinnitus loudness (in decibel) assessed by loudness matching test | Change in tinnitus loudness was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in Tinnitus loudness at three months assessed by Loudness matching audiometric test
Tinnitus Handicap Inventory Questionnaire score (ranging from 0 to 100) which assesses the impact of tinnitus on daily life | Change in Tinnitus Handicap Inventory score was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in Tinnitus Handicap Inventory Questionnaire at three months

SECONDARY OUTCOMES:
Tinnitus frequency (in Hz) assessed by pitch match test | Change in Tinnitus frequency was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in Tinnitus frequency at three months
Tinnitus Functional Index questionnaire score (ranging from 0 to 100) which assesses the impact of tinnitus on daily life | Change in Tinnitus Functional Index score was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in Tinnitus Functional Index score at three months
serum Total Antioxidant Capacity (mM) | Change in Serum Total Antioxidant Capacity was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in Serum Total Antioxidant Capacity at three months
Vitamins B12, E, C, B2, B1, B6 and folic acid in blood | Change in vitamin levels were assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in vitamin levels at three months
Tinnitus Minimum Masking Level (in decibel) | Change in Tinnitus Minimum Masking Level was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in Tinnitus Minimum Masking Level at three months
Visual Analogue Scale Score (ranging from 0 to 10) which assesses tinnitus annoyance | Change in Visual Analogue Scale Score was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in Visual Analogue Scale Score at three months
serum Superoxide Dismutase (U/ml) | Change in serum Superoxide Dismutase was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in serum Superoxide Dismutase at three months
serum Oxidized LDL (ng/ml) | Change in serum Oxidized LDL was assessed at 3 months from baseline in tinnitus patients
  Mean Change from Baseline in serum Oxidized LDL at three months

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Xenelis, Professor, Study Director — General Hospital of Athens "Hippocratio", Department of Otorhinolaryngology
Locations (1):
- General Hospital of Athens "Hippocratio", Department of Otorhinolaryngology, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided